CLINICAL TRIAL: NCT02402049
Title: Is Homeopathic Treatment a Placebo Treatment? - Homeopathic Treatment of Premenstrual Syndrome- A Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Homeopathic Treatment of Premenstrual Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMS-14
Record Dates: First submitted 2015-03-12; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Premenstrual Syndrome-PMS
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- 1: Natrum muriaticum 30C (Active Comparator): Natrum muriaticum 30C
  Interventions: Drug: Natrum muriaticum 30C
- 2: Lachesis 30C (Active Comparator): Lachesis 30C
  Interventions: Drug: Lachesis 30C
- 3: Sepia 30C (Active Comparator): Sepia 30C
  Interventions: Drug: Sepia 30C
- 4: Nux vomica 30C (Active Comparator): Nux vomica 30C
  Interventions: Drug: Nux vomica 30C
- 5: Pulsatilla 30C (Active Comparator): Pulsatilla 30C
  Interventions: Drug: Pulsatilla 30C
- 6 Folliculinum 30C (Active Comparator): Folliculinum 30C
  Interventions: Drug: Folliculinum 30C
- 1: Placebo Natrum muriaticum (Placebo Comparator): Placebo Natrum muriaticum
  Interventions: Drug: Placebo Natrum muriaticum
- 2: Placebo Lachesis (Placebo Comparator): Placebo Lachesis
  Interventions: Drug: Placebo Lachesis
- 3: Placebo Sepia (Placebo Comparator): Placebo Sepia
  Interventions: Drug: Placebo Sepia
- 4: Placebo Nux vomica (Placebo Comparator): Placebo Nux vomica
  Interventions: Drug: Placebo Nux vomica
- 5: Placebo pulsatilla (Placebo Comparator): Placebo pulsatilla
  Interventions: Drug: Placebo pulsatilla
- 6: Placebo Folliculinum (Placebo Comparator): Placebo Folliculinum
  Interventions: Drug: Placebo Folliculinum

INTERVENTIONS:
Drug: Natrum muriaticum 30C — 3 globules of Natrum muriaticum applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Natrum muriaticum
  Arms: 1: Natrum muriaticum 30C
Drug: Lachesis 30C — 3 globules of Lachesis applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Lachesis
  Arms: 2: Lachesis 30C
Drug: Sepia 30C — 3 globules of Sepia applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Sepia
  Arms: 3: Sepia 30C
Drug: Nux vomica 30C — 3 globules of Nux vomica applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Nux vomica
  Arms: 4: Nux vomica 30C
Drug: Pulsatilla 30C — 3 globules of Pulsatilla applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Pulsatilla
  Arms: 5: Pulsatilla 30C
Drug: Folliculinum 30C — 3 globules of Folliculinum applied once daily at days 7,8, and 9 after the start of the period.
  Other Names: Active Folliculinum
  Arms: 6 Folliculinum 30C
Drug: Placebo Natrum muriaticum — 3 globules of placebo Natrum muriaticum applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 1: Placebo Natrum muriaticum
Drug: Placebo Lachesis — 3 globules of placebo Lachesis applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 2: Placebo Lachesis
Drug: Placebo Sepia — 3 globules of placebo Sepia applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 3: Placebo Sepia
Drug: Placebo Nux vomica — 3 globules of placebo Nux vomica applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 4: Placebo Nux vomica
Drug: Placebo pulsatilla — 3 globules of placebo Pulsatilla applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 5: Placebo pulsatilla
Drug: Placebo Folliculinum — 3 globules of placebo Folliculinum applied once daily at days 7,8, and 9 after the start of the period.
  Arms: 6: Placebo Folliculinum

SUMMARY:
The proposed study will focus on premenstrual syndrome (PMS) symptom alleviation for women diagnosed as suffering from the syndrome with the DRSP questionnaire.

The women will be treated with Homeopatic remedies. The improvement of PMS symptoms will be evaluated using the Daily Record of Severity of Problems questionnaire (DRSP). The questionnaire will be completed daily by women for 2 months prior to receiving the treatment and for 3 months following treatment with a single dose of the homeopathy treatment.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is a set of physical, emotional and behavioral symptoms that occur during the week preceding menstruation and which alleviate when the menstrual flow begins. PMS affects millions of women during their reproductive years. Mild symptoms, which usually do not interfere with daily activities, are experienced occasionally by almost all ovulatory women. Between 8-30% of ovulatory women suffer from moderate to severe PMS symptoms, which may even require treatment. The more severe form of PMS, premenstrual dysphoric disorder is considered to affect up to 8% of ovulatory women. This severe form is associated with severe disruptions in work function, family, or social relationships. To date, therapeutic interventions are insufficient and ranges from stress reduction and lifestyle changing to hormonal therapies and the use of psychotropic medications. While traditional medications do not necessarily offer satisfactory alleviation of PMS symptoms homeopathy can offer a significant alleviation of PMS symptoms for an extended period of time.

The proposed study will focus on PMS symptom alleviation for women diagnosed as suffering from the syndrome with the DRSP questionnaire.

Five Homeopathic remedies (Natrum muriaticum, Lachesis, Sepia, Nux vomica and Pulsatilla ) will be used, in five different therapy groups. The women will be allocated to the groups according to their matching to the remedy according to Homeopathic principles. In each group the women will either be treated with the appropriate remedy or with a placebo remedy. Women who do not match any of these five groups will be allocated to a sixth group receiving either Folliculinum that is given as general indication for PMS in homeopathy or placebo.

The improvement of PMS symptoms will be evaluated using the Daily Record of Severity of Problems questionnaire at (DRSP). The questionnaire will be completed daily by women for 2 months prior to receiving the treatment and for 3 months following treatment with a single dose of the homeopathy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Suffers from the PMS, confirmed by the DRSP questionnaire, for at least one year
* Read and write in
* Signing the informed consent form

Exclusion Criteria:

* Comorbidity.
* Use of medications.
* Menstruation complains which do not correlate to the menstruation cycle.
* Inability to be in a daily contact with the experiment center (e.g., by phone, electronically).
* Participating in another clinical trial in the last 30 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Decrease in the average DRSP questionnaire scores during the 12 days prior to menstruation during three months following single dose homeopathy treatment as compared to the average DRSP questionnaire scores during the 12 days prior to menstruation during | 3 months

SECONDARY OUTCOMES:
Decreased work absence during the 3 months after therapy begin as compared to the 2 months prior to homeopathy treatment. | 3 months
Change in the amount of painkillers taken by the patient during the 3 months after homeopathy treatment as compared to the amount of medications taken by the patient during 2 months prior to therapy begin. | 3 months
Self-report of the efficiency of the homeopathy treatment. | 3 months
  The patient will indicate subjectivlly her filling after taking the homeopathic remedy
Side effects occurrence during therapy (e.g headaches, vomiting, nausea etc.) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — The Center for Inegrative Complementary Medicine, Shaare Zedek Medical Center, Jerusalem, Israel